CLINICAL TRIAL: NCT01864395
Title: Clinical and Chemical Outcomes Following Cardiac Surgery: The Post-Operative Effects of Modified Ultrafiltration (On-line MUF) and Off-line (MUF)
Brief Title: Clinical and Chemical Outcomes Following Cardiac Surgery: The Post-Operative Effects of MUF
Acronym: MUF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-143
Record Dates: First submitted 2013-05-14; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease; Anemia
Keywords: cardiovascular surgery; cardiac surgery; cardiopulmonary bypass; IV fluids; blood pressure; heart-lung machine; hemofilter; online MUF; offline MUF; modified ultrafiltration; multiple-pass hemofiltration; centrifugation method; blood transfusion; plasma proteins; post-cardiopulmonary bypass; hemoglobin; clotting factors; systemic blood pressure; cardiac index; cytokines; post-operative bleeding; protamine administration; patient size; allogeneic transfusion; total protein; albumin; vasoactive inotrope score; fluid balance; chest tube loss; length of stay; ventilation time; markers of inflammation
MeSH Terms: conditions — Coronary Artery Disease; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (CF) (Experimental): Centrifugation Method (CF): currently used to separate whole blood into red blood cells (RBCs) and plasma components. The RBCs are washed with normal saline and re-infused into the patient, while the plasma portion is discarded.
  Interventions: Procedure: Centrifugation Method
- Online MUF (Experimental): Online MUF: hemofilter is used online while the heart-lung machine is connected to the patient.
  Interventions: Procedure: Online MUF
- Offline MUF (Experimental): Offline MUF: hemofilter is used offline when the heart-lung machine is not connected to the patient.
  Interventions: Procedure: Offline MUF

INTERVENTIONS:
Procedure: Centrifugation Method — Currently used to separate whole blood into red blood cells (RBCs) and plasma components. The RBCs are washed with normal saline and re-infused into the patient, while the plasma portion is discarded.
  Arms: Control (CF)
Procedure: Online MUF — Hemofilter is used online while the heart-lung machine is connected to the patient.
  Arms: Online MUF
Procedure: Offline MUF — Hemofilter is used offline when the heart-lung machine is not connected to the patient.
  Arms: Offline MUF

SUMMARY:
It is hypothesized that on-line modified ultrafiltration (MUFF) post-cardiopulmonary bypass will result in improved patient outcomes over the 12-hour post-operative period as compared to control and off-line MUFF.

DETAILED DESCRIPTION:
Current practice in cardiac surgery requiring cardiopulmonary bypass (CPB) dictates the salvage of the residual circuit volume at the end of the procedure into an autologous recovery system. This system uses the centrifugation method (CF) to separate whole blood into red blood cells (RBCs) and plasma components (Sutton et al, 1993). The RBCs are then washed with normal saline and re-infused into the patient as needed while the plasma components are discarded.

While this technique produces a product with a high haemoglobin (Hb), the main disadvantage of this process is the loss of plasma protein and clotting factors (Samolyk et al, 2005).

The Modified Ultrafitration (MUF) is a standard of care technique that was originally used on pediatric patients undergoing cardiac surgery with CPB. Following CPB while the aorta is still cannulated, MUF uses an inline hemofilter to concentrate the patients total blood volume thereby increasing Hb, plasma proteins, systemic blood pressure, and cardiac index while decreasing cytokines and post-operative bleeding (Kiziltepe et al. 2001).

According to a task-force on evidence based surgery (the Society of Thoracic Surgeons and the Society of Cardiovascular Anesthesia) the use of modified ultrafiltration (online-MUF) is indicated for blood conservation and reduction of post-operative blood loss in adult cardiac operations using cardiopulmonary bypass (CPB) (Ferraris et al 2011). Moreover, Luciani et al. 2001, showed significantly lower levels of GI, neurologic and cardiac complications in patients who underwent on-line MUF following cardiac surgery as compared to those who did not. They also demonstrated a significantly lower mortality at 30 days follow-up in patients receiving online MUF as compared to control. Boodhwani et al. (2006) demonstrated that the use of online MUF was associated with a 0.72 unit reduction in blood transfused and a reduction of post-operative loss. The disadvantages to this technique are the time required (10-15 min), delays protamine administration, and the requirement of anaesthesia cooperation for pressure management. According to the Proceedings of the American Society of Extracorporeal Technology International Conf. March 9, 2013, online MUF works best and is recommended for smaller patients 75 kg or less because the effect of concentration of the blood volume is greater in smaller patients as compared to larger patients. In house data collected by our Department of Clinical Perfusion at the Royal University Hospital has demonstrated that 70% of the smaller patients undergoing cardiac surgery (mainly women) receive allogeneic transfusion peri- and post-operatively.

Off-line MUFF, another standard of care technique, is used after separation from CPB and decannulation. This technique uses a hemofilter to concentrate the residual CPB volume to produce a product which is more analogous to whole blood as compared to that processed by the CF method. Recently, our research group has shown that after 12-hours post-operatively patients' biochemical (total protein and albumin) and clinical parameters (vasoactive inotrope score and fluid balance) were significantly improved when patients' residual CPB volume underwent multiple-pass hemofiltration as compared to the CF (McNair et al. (2013), Journal of Cardiothoracic and Vascular Anaesthesia, In Press). Recently, it has been demonstrated that following cardiac surgery, the post-operative use of vasoactive inotropes is decreased when the residual CPB volume is processed by the offline MUF method as compared to the CF method (Coli et al 2012; McNair et al. (2013), Journal of Cardiothoracic and Vascular Anaesthesia, In Press). The disadvantages of on-line MUFF are the possible entrainment of air into the arterial line and prolonged time for protamine administration. The disadvantages of off-line MUFF are inadequate clearance of heparin by the hemofilter and prolonged processing time.

There is a need for the proposed study because it will help to determine whether there is any difference in patient outcomes between the use of on-line MUF and off-line MUF. Our study will also demonstrate which method is better at enhancing clinical (volume of allogeneic transfusion, chest tube loss, fluid balance length of stay and ventilation time) and biochemical (Hb, total protein, albumin and markers of inflammation) outcomes during the 12-hour post-operative period.

The data gathered from this study may save smaller patients from exposure to allogeneic transfusions during the 12-hour postoperative period. This study will also determine which method our institution will use to better serve our patients, allowing them to have a safer, shorter, transfusion-free recovery during the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* patient weighs 75 kg or smaller
* 40-80 years of age
* elective or urgent cardiac surgery

Exclusion Criteria:

* emergent surgery
* severe anemia
* severe kidney dysfunction
* ejection fraction of less than 30%

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Volume of Chest Tube Drainage | 12 hours
  Our primary outcome variable is the post-operative volume of chest tube drainage.

SECONDARY OUTCOMES:
Biochemical Variables | 12 hours
  Biochemical variables include Hb, albumin fibrinogen, and total protein.
Clinical Variables | 12 hours
  Clinical variables include volume of allogeneic transfusion, length of stay in ICU, intubation time, and vasoactive inotrope score.

CONTACTS AND LOCATIONS:
Overall Officials: Erick D McNair, PhD, Principal Investigator — Clinical Assistant Professor, Department of Surgery, Cardiovascular Surgery
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada